CLINICAL TRIAL: NCT03157453
Title: Comparison of Two Initial Evaluation Scales of the Severity of Brain Injury Adults
Brief Title: Comparison of Two Initial Evaluation Scales of the Severity of Brain Injury Adults Patients on the Neurological Outcome at 6 Months
Acronym: CASSANDRA
Status: Terminated | Type: Observational
Why Stopped: Recruitment difficulty
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CASSANDRA
Record Dates: First submitted 2017-03-17; First posted 2017-05-17 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Brain Injury
Keywords: Evaluation scale; Brain injury; Severity of Brain Injury; Initial Evaluation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective cohort study. Any patient with potential cerebral injured (medical or traumatic) will be included in the study, regardless of its severity, history, the presence of anticoagulant or antiagrégant.

The collection should be done as soon as possible, in the reception of vital emergencies or in the urgencies. The collection consists of the realization of a Glasgow score and a scale of Kremlin-Bicêtre for all patients by completing a standardized collection sheet. The collection of GCS and Kremlin-Bicêtre must be did at the same time. The collection sheet is filled by medical personnel trained.

The future of the patient is informed at 6 months using the Glasgow Outcome Scale- Extended, which will be made during a following consultation or by phone. Additional data will be collected on the folder (ventilation time, days of hospitalization, mortality).

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or more
* Potentially Victim of a cerebral injury whatever the level of severity
* Having a calculation of GCS and KBS on arrival at the hospital (emergency room)
* Affiliated to a social security scheme or benefiting through a third person.

Exclusion Criteria:

* Pregnant women
* Patients who refusing to participate in research
* Patients undergoing enhanced protection (persons deprived of liberty by a judicial or administrative decision, adults under legal protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with potential cerebral injured (medical or traumatic) will be included in the study, regardless of its severity, history, the presence of anticoagulant or antiagrégant.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Comparison of ROC curve areas of the two scales to predict an unfavorable neurological prognosis at 6 months (GOS-E < or = 5) | 6 months

SECONDARY OUTCOMES:
Comparison of ROC curve areas of the two scales to predict an unfavorable neurological prognosis at 6 months (GOS-E < or = 5) for medical injury | 6 months
Comparison of ROC curve areas of the two scales to predict an unfavorable neurological prognosis at 6 months (GOS-E < or = 5) for traumatized cranial | 6 months
Mortality in intensive care unit | 6 months
Duration of stay in intensive care unit | 6 months
Duration of mechanical ventilation | 6 months
Mortality at hospital | 6 months
Mortalit at 6 months | 6 months
Duration of stay at hospital | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Poitiers, Poitiers, France